CLINICAL TRIAL: NCT01410214
Title: A Phase II Trial of Erlotinib Versus Combination of Vinorelbine Plus Cisplatin as Adjuvant Treatment in Stage IIIA Non-small-cell Lung Cancer After Complete Resection With Sensitizing EGFR Mutation in Exon 19 or 21 and Wild-type K-ras
Brief Title: Erlotinib Versus Vinorelbine/Cisplatin as Adjuvant Treatment in Stage IIIA NSCLC Patients With EGFR Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Lung Cancer Surgical Group (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Fudan University (Other); Zhejiang Cancer Hospital (Other); Peking University Cancer Hospital & Institute (Other); Sun Yat-sen University (Other); Chinese PLA General Hospital (Other); Qingdao University (Other); The First Affiliated Hospital of Soochow University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Hebei Medical University Fourth Hospital (Other); The Second People's Hospital of Sichuan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-LCSG-001
Record Dates: First submitted 2011-08-01; First posted 2011-08-05 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Non-small Cell Lung Cancer Stage IIIA
Keywords: NSCLC; EGFR Mutation Positive; complete resection; Erlotinib Versus NVB/Cisplatin as Adjuvant treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Vinorelbine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erlotinib arm (Experimental): In the adjuvant treatment phase, erlotinib 150 mg/day taken orally for 2 years or till disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib
- Chemo arm (Active Comparator): In the adjuvant treatment phase, patient will receive vinorelbine 25mg/m2 IV on day 1 and day 8, and cisplatin 25mg/m2 on day 1 and day 2 and day 3, of a 3-week schedule for 4 cycles or till disease progression or unacceptable toxicity.
  Interventions: Drug: vinorelbine/cisplatin

INTERVENTIONS:
Drug: Erlotinib — In the adjuvant treatment phase, erlotinib 150 mg/day taken orally for 2 years or till disease progression or unacceptable toxicity.
  Other Names: tarceva
  Arms: Erlotinib arm
Drug: vinorelbine/cisplatin — In the adjuvant treatment phase, patient will receive vinorelbine 25mg/m2 IV on day 1 and day 8, and cisplatin 25mg/m2 on day 1 and day 2 and day 3, of a 3-week schedule for 4 cycles or till disease progression or unacceptable toxicity.
  Other Names: NP; NVB/cisplatin
  Arms: Chemo arm

SUMMARY:
The purpose of this study is to assess the effect and safety of erlotinib versus NVB plus cisplatin (NP) as adjuvant treatment in patients with stage IIIA NSCLC after complete resection with EGFR activating mutations and to explore a new treatment strategy for this subset.

DETAILED DESCRIPTION:
The LACE meta-analysis identified four cycles of platinum-based program to improve II~IIIA stage completely resected NSCLC pts the role of 5-year survival, but its treatment-related life threatening toxicity limits its use. The EGFR tyrosine kinase inhibitor (TKI) may provide a dramatic response in pts with pulmonary adenocarcinoma carrying EGFR activating mutations in the metastatic setting. The aim of this study is to investigate the efficacy and safety of erlotinib versus NVB plus cisplatin (NP) as adjuvant treatment in pts with stage IIIA NSCLC after Complete Resection with EGFR activating mutations and to explore a new treatment strategy for this subset.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Males or females aged ≥18 years.
* Chest CT, brain CT or MRI, ECT, abdominal and double-neck B-, or whole body PET-CT examination in 4 weeks before complete resection.
* Pathological diagnosed of non-small cell lung cancer.
* Diagnosed as stage IIIA.
* In 4 weeks after complete resection pts start to accept the adjuvant therapy in this study, previously did not receive any anti-tumor therapy.
* EGFR activating mutation in exon 19 or 21 and KARS
* ECOG performance status 0-1.
* Life expectancy ≥3 months.
* Adequate hematological function:Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN);Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN.
* Adequate renal function:Serum creatinine ≤ 1.25 x ULN, and creatinine clearance ≥ 60 ml/min.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Patients must be nonpregnant and non-lactating.Patients of childbearing potential must implement an effective method of contraception during the study. All female Patients, except those who are postmenopausal or surgically sterilized, must have a negative pre-study serum or urine pregnancy test. .

Exclusion Criteria:

* Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
* Patients with prior chemotherapy or therapy with systemic anti-tumour therapy.
* Patients with prior radiotherapy.
* History of another malignancy in the last 5 years with the exception of the following:Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Any evidence confirmed tumor recurrence before adjuvant treatment.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Any evidence of clinically active interstitial lung disease.
* Eye inflammation or eye infection not fully treated or conditions predisposing the subject to this.
* Known human immunodeficiency virus (HIV) infection.
* Known hypersensitivity to Tarceva or NVB or cisplatin.
* Pregnancy or breast-feeding women.
* ECOG performance status ≥ 2.
* Ingredients mixed with small cell lung cancer patients
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or puts the subject at high risk for treatment-related complications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  To evaluate Disease-free survival(DFS) of two groups

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 2 years
  To evaluate the safety profile(Number of Participants with Adverse Events) of two group.
Quality of Life (QOL) | 2 years
  To evaluate the Quality of Life (QOL) of two group.
overall survival (OS) | 2 years
  To evaluate the overall survival (OS) of two groups

CONTACTS AND LOCATIONS:
Overall Officials: Changli Wang, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (11):
- China (11):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiurted Hospital of Soochow University, Suzhou, Jiangsu
  - Qingdao University Medical College, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The Second People's Hospital of Sichuan, Chengdu, Sichuang
  - Tianjin Medical University Cancer Institute and Hospital, Tianji, Tianji
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang